CLINICAL TRIAL: NCT07134179
Title: Insufficient Regional Anesthesia for Cesarean Section: Mothers' Experiences A Qualitative Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Helene Korvenius Nedergaard, MD, associate professor, Sygehus Lillebaelt
Other Study IDs: REC607
Record Dates: First submitted 2025-07-08; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Caesarean Section; Regional Anesthesia
Keywords: pain during caesarean section; insufficient regional anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women, who experienced pain during caesarean delivery: Adult women, who underwent elective or emergency cesarean delivery within the last 2 years, with the experience of pain during surgery, under regional (spinal or epidural or combined epidural-spinal) anesthesia, that was not converted to general anesthesia
  Interventions: Other: Experience of pain during caesarean delivery

INTERVENTIONS:
Other: Experience of pain during caesarean delivery — We wish to investigate how women experience insufficient regional anesthesia during cesarean sections, in cases where the regional anesthesia was not converted to general anesthesia. The focus is on exploring the factors that contribute positively and negatively to the woman's experience in this situation

SUMMARY:
In Denmark, approximately 20% of all children are born via cesarean section (C-section), making it the most common surgical procedure (also internationally). The recommended anesthesia for cesarean sections is regional anesthesia (spinal or epidural, "spinal anesthesia"), as it has several advantages: the woman is awake and experiences the delivery of her child, she maintains spontaneous breathing. Furthermore, regional anesthesia can contribute to early postoperative pain management to some extent.

With spinal anesthesia, most women feel pressure and touch but no pain during the cesarean section. However, some women do experience pain during the procedure, necessitating further intervention or ultimately a change in anesthetic form. If inadequate anesthesia is detected before the surgery begins, one may choose to administer renewed regional anesthesia (typically an epidural). However, if the woman first experiences pain after the surgery has commenced, it can be necessary to place her under general anesthesia for the remainder of the procedure. Experience shows that this process can be challenging, and there are frequent examples in clinical practice of inappropriate courses of action, where women have experienced unacceptable pain during their cesarean sections without being placed under general anesthesia.

The consequences of inadequate anesthesia for cesarean sections can be quite significant for women, including impaired bonding with the child, poorer establishment of breastfeeding, increased risk of postpartum reactions and post-traumatic stress.

The aim of this study is to investigate how women experience insufficient regional anesthesia during cesarean sections, in cases where the regional anesthesia was not converted to general anesthesia. The focus is on exploring the factors that contribute positively and negatively to the woman's experience in this situation, and investigate if any recommendations for how to handle the situation can be extrapolated from the women's experiences.

Method Qualitative study.

Inclusion criteria:

* Adult women undergoing elective or emergency cesarean delivery within the last 2 years, with the experience of pain during surgery
* Regional (spinal or epidural or combined epidural-spinal) anesthesia NOT converted to general anesthesia

Exclusion criteria:

* Does not speak Danish or English
* Does not wish to participate

Relevant women will be invited to contact us through public post on social media. If a woman responds to the post, she will be offered further information about the project, both verbally via telephone and in writing sent by email.

Women can also be invited to participate if encountered by a project-group member during clinical work.

Participants will be invited to an interview via telephone. This will take place as a semi-structured interview, initiated with open questions and concluded with a few more specific questions. At the end of the interview, a screening for post-traumatic stress will be conducted using the PTSD-8 tool.

Interviews will be recorded digitally and transcribed verbatim. The interview guide will be developed with input from the entire project group and with participation from three mothers who have previously experienced insufficient regional anesthesia during a cesarean section. The guide will be pilot-tested on 2-3 patients after cesarean section. The interview guide may be adjusted during the study, if necessary.

The number of women required to participate before a sufficient amount of information is obtained (as no new information is expected from subsequent interviews) is not known in advance; however, it is estimated that 20 women will need to participate. However, the sample size is also defined by convenience, as the investigators do not know how many women it will be possible to establish contact with via the Facebook post and through clinical work. If too few women (e.g. <15) are included within the first two months, the investigators will make a new public posting and expand the period of inclusion to concern cesarean sections within the last 5 years instead of 2 years.

Baseline data regarding the mother and the cesarean section will be collected by asking the women during the scheduled interview, and therefore access to medical records are not necessary. Qualitative data will also be gathered through the interview, conducted as a semi-structured interview based on an interview guide.

Data will be entered into SurveyXact software, where it will be securely stored. Data will be handled using descriptive statistics. Interview data will be analyzed using content analysis. Nvivo software will be used for managing and coding qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective or emergency cesarean delivery within the last 2 years, with the experience of pain during surgery
* Regional (spinal or epidural or combined epidural-spinal) anesthesia NOT converted to general anesthesia
* Age ≥18 years

Exclusion Criteria:

* Does not speak Danish or English
* Does not wish to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women, who have undergone elective or emergency caesarean delivery within the past 2 years under regnional anesthesia and experienced pain during the operation without conversion to general anesthesia will be invited to participate, either via posts on social media or when met in clinical work.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Experience of pain during caesarean section | Experience of caesarean delivery, max 2 years ago
  The primary outcome is the women's experience of pain during caesarean delivery. This will be assessed through the qualitative method "manifest content analysis". All participating women will be interviewed using a semi-structured model based on an interview guide. All interviews will be transscribed verbatim and analysed by three to four researchers to identify relevant themes, describing the women's experience.

SECONDARY OUTCOMES:
Posttraumatic stress | Posttraumatic stress related to caesarean delivery max 2 years ago
  Screening for posttraumatic stress, using the PTSD-8 inventory (in Danish), verbally during the telephone interview. The PTSD-8 inventory consists of 8 questions regarding the event (in this case the cesarean section). Each question can be answered with "not at all, rarely, sometimes of often", which corresponds to 1, 2, 3 and 4 points, respectively. Total score will be between 0 and 32. Higher scores indicates higher likelyhood of posttraumatic stress.

IPD SHARING:
Plan to Share IPD: No
IPD in this study will be confidential interviews.